CLINICAL TRIAL: NCT00127218
Title: HDL Increased Plaque Stabilization in the Elderly
Brief Title: High-Density Lipoprotein (HDL) Cholesterol Increased Plaque Stabilization in the Elderly
Acronym: NIA-Plaque
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00035188; 5R01AG021570-03 (NIH)
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Atherosclerosis; Cardiovascular Disease
Keywords: atherosclerotic plaque; MRI; inflammatory markers; statins
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Plaque, Atherosclerotic | interventions — Fluvastatin; Pravastatin; Simvastatin; Ezetimibe, Simvastatin Drug Combination; Atorvastatin; Rosuvastatin Calcium; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): any statin plus niacin
  Interventions: Drug: any statin; Drug: niacin
- 2 (Placebo Comparator): any statin plus placebo
  Interventions: Drug: any statin; Drug: Placebo

INTERVENTIONS:
Drug: any statin — Participants will be provided a prescription for fluvastatin 80 mg to be taken on a daily basis, or they may continue their ongoing or any other cholesterol-lowering drugs such as pravastatin 80 mg daily, simvastatin 20 mg daily, atorvastatin up to 20 mg daily or rosuvastatin up to 20 mg daily for 18 months
  Other Names: fluvastatin (Lescol); pravastatin (Pravachol); simvastatin (Vytorin); atorvastatin (Lipitor); rosuvastatin (Crestor)
Drug: niacin — long-acting niacin daily for 18 months
  Arms: 1
Drug: Placebo — matching placebo pill daily for 18 months
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the added benefits of increased high-density lipoprotein (HDL) cholesterol serum levels over and above those achieved by lipid lowering therapy guided by current guidelines, in older individuals with cardiovascular disease.

DETAILED DESCRIPTION:
The hypothesis being tested is that the current standard lipid lowering therapy, combined with a 20 percent or greater increase in serum HDL induced by long-acting niacin, reduces plaque size in older individuals with cardiovascular disease. The specific aims of testing this hypothesis are:

1. to determine the effects of statin plus placebo vs. statin plus niacin therapy on plaque size and composition,
2. to determine whether alterations of inflammatory markers of atherosclerosis induced by lipid lowering therapy parallel alterations of plaque architecture and composition in older patients with cardiovascular disease,
3. to determine the effects of these interventions on the incidence of cardiovascular and cerebrovascular events.

The results of the trial will be directly applicable to developing strategies for plaque stabilization in the elderly who suffer the most from the severe complications of advanced cardiovascular atherosclerosis.

A total of 144 participants aged 65 and older with cardiovascular or cerebrovascular disease will be recruited. Participants will be randomized to receive either statin plus niacin or statin plus a placebo for 18 months. Participants will be provided a prescription for fluvastatin 80 mg to be taken on a daily basis, or they may continue their ongoing or any other cholesterol-lowering drugs such as pravastatin 80 mg daily, simvastatin 20 mg daily, atorvastatin up to 20 mg daily or rosuvastatin up to 20 mg daily. Ten visits are expected, initially every 4 weeks for dose adjustment. Then visits will be every 6 months; MRI, Inflammatory Markers tests, and other lab tests will be done at baseline and the visits at months 6, 12, and 18.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* Documented clinical cardiovascular or cerebrovascular disease due to atherosclerosis
* Candidate for lipid lowering therapy; no contraindication to fluvastatin, niacin or aspirin therapy
* Low-density lipoprotein (LDL) cholesterol below 150 mg/dl if untreated or below 125 mg/dl on statin monotherapy
* Willing to discontinue present therapy if private physician agrees with enrollment
* Eligible to undergo trans-esophageal magnetic resonance imaging (MRI); no contraindications to Gadolinium-DTPA, the contrast agent used
* Willing to sign Informed Consent

Exclusion Criteria:

* Ineligibility for MRI procedure due to pacemaker, metal implants, or other ferromagnetic devices
* Claustrophobia
* Previously documented esophageal disease which would preclude trans-esophageal MRI
* LDL-C greater than 150 mg/dl off lipid lowering therapy or daily statin therapy requiring doses greater than 20 mg of atorvastatin, 20 mg of simvastatin, 80 mg of lovastatin, 80 mg of pravastatin, 80 mg of extended release fluvastatin, or 20 mg of rosuvastatin
* Contraindication or allergy to statins or aspirin
* Current use of or known intolerance or allergy to Niaspan (a long-acting niacin)
* Allergy or intolerance to Gadolinium-DTPA (MRI contrast agent)
* Liver or kidney failure defined clinically and by laboratory data
* Mental, neurologic or social condition preventing understanding of the rationale, procedures, risks and potential benefits associated with the trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 145 (Actual)
Dates: Start 2003-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Unversity School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Guyton JR, Goldberg AC, Kreisberg RA, Sprecher DL, Superko HR, O'Connor CM. Effectiveness of once-nightly dosing of extended-release niacin alone and in combination for hypercholesterolemia. Am J Cardiol. 1998 Sep 15;82(6):737-43. doi: 10.1016/s0002-9149(98)00448-2. PMID 9761083
- [Background] Ballantyne CM, Herd JA, Ferlic LL, Dunn JK, Farmer JA, Jones PH, Schein JR, Gotto AM Jr. Influence of low HDL on progression of coronary artery disease and response to fluvastatin therapy. Circulation. 1999 Feb 16;99(6):736-43. doi: 10.1161/01.cir.99.6.736. PMID 9989957
- [Background] Brown BG, Zhao XQ, Chait A, Fisher LD, Cheung MC, Morse JS, Dowdy AA, Marino EK, Bolson EL, Alaupovic P, Frohlich J, Albers JJ. Simvastatin and niacin, antioxidant vitamins, or the combination for the prevention of coronary disease. N Engl J Med. 2001 Nov 29;345(22):1583-92. doi: 10.1056/NEJMoa011090. PMID 11757504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 1:1 ratio to receive niacin or placebo, using a random number schema stratiﬁed to ensure equal numbers between age 65-74 years and 75 years and above. Study took place in a university outpatient center.
Pre-assignment Details: Participants were over age 65 years with a history of cardiovascular events or evidence of atherosclerosis at angiography (>50% stenosis) or non-invasive imaging, with baseline LDL<3.24 mmol/L if already on statin therapy and <3.89 mmol/L if untreated. There were no restrictions on HDL level.
Groups:
- Niacin Plus Statin: Extended release niacin (1500 mg daily) plus statin therapy to reach their National Cholesterol Education Program-deﬁned low density lipoprotein (LDL)cholesterol target
- Placebo Plus Statin: placebo plus statin therapy to reach their National Cholesterol Education Program-deﬁned low density lipoprotein (LDL)cholesterol target
Period: Overall Study
Arm/Group | Niacin Plus Statin | Placebo Plus Statin
Started | 72 | 73
Completed | 59 | 58
Not Completed | 13 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin Plus Statin | Placebo Plus Statin | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [69 to 77] | 72 [69 to 77] | 73 [69 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 58 | 60 | 118
Region of Enrollment [Number; unit: participants]
  United States | 72 | 73 | 145

OUTCOME MEASURES:

1. Primary Outcome: Changes in Plaque Architecture and Composition Directly Measured by Magnetic Resonance Imaging (MRI) in the Aorta and Carotid Arteries
Description: The primary endpoint is Changes in plaque architecture and composition directly measured by magnetic resonance imaging (MRI) in the aorta and carotid arteries.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: percentage of internal carotid artery
Arm/Group | Niacin Plus Statin | Placebo Plus Statin
Number analyzed (Participants) | 72 | 73
percentage of internal carotid artery | 7 (.2) | 5 (.2)

2. Secondary Outcome: Multiple Combined Events ( Cardiovascular and Cerebrovascular Events as Well as Myocardial Revascularization)
Description: Cerebrovascular events (newly diagnosed) such as Stroke and Myocardial revascularization (specifically coronary artery bypass grafting, percutaneous coronary interventions, carotid endarterectomy) were recorded
Time Frame: 18 months
Population: Cardiovascular event (stroke) was seen in only 1 patient and 5 patients needed myocardial revascularization
Measure: Count of Participants; unit: Participants
Groups:
- Any Statin Plus Niacin: any statin plus niacin
  any statin: Participants will be provided a prescription for fluvastatin 80 mg to be taken on a daily basis, or they may continue their ongoing or any other cholesterol-lowering drugs such as pravastatin 80 mg daily, simvastatin 20 mg daily, atorvastatin up to 20 mg daily or rosuvastatin up to 20 mg daily for 18 months
  niacin: long-acting niacin daily for 18 months
- Any Statin Plus Placebo: any statin plus placebo
  any statin: Participants will be provided a prescription for fluvastatin 80 mg to be taken on a daily basis, or they may continue their ongoing or any other cholesterol-lowering drugs such as pravastatin 80 mg daily, simvastatin 20 mg daily, atorvastatin up to 20 mg daily or rosuvastatin up to 20 mg daily for 18 months
  Placebo: matching placebo pill daily for 18 months
Arm/Group | Any Statin Plus Niacin | Any Statin Plus Placebo
Number analyzed (Participants) | 72 | 73
Participants | 6 | 2

ADVERSE EVENTS:
Arm/Group | Niacin Plus Statin | Placebo Plus Statin
Serious Adverse Events (participants affected / at risk) | 1/72 | 1/73
Other Adverse Events (participants affected / at risk) | 5/72 | 2/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin Plus Statin (N=72) | Placebo Plus Statin (N=73)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Death (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin Plus Statin (N=72) | Placebo Plus Statin (N=73)
Coronary Revascularization (Vascular disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No